CLINICAL TRIAL: NCT03401645
Title: Home-based Arm and Hand Exercise (HAHE) to Improve Upper Limb Function After Traumatic Brain Injury
Brief Title: Home-based Arm and Hand Exercise to Improve Upper Limb Function After Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Peii Chen, Senior Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-974-17
Record Dates: First submitted 2018-01-02; First posted 2018-01-17 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Alarm Active) (Experimental): Participants will be wearing the wrist device with an alarm timer that sends out signals every 5 minutes. The alarm is a buzzing noise and a vibration. Participants must turn off the alarm then perform a series of visuomotor tasks. This will be done for one hour, twice a day for two weeks.
  Intervention: Device - Wrist Alarm; Behavioral - Home-based Arm and Hand Exercise
  Interventions: Other: Wrist Alarm; Behavioral: Home-based Arm and Hand Exercise
- Control (Sham Control) (Sham Comparator): Participants will perform the same tasks as the Alarm/Treatment group, but without the alarm timer. This is a series of visuomotor tasks for one hour, twice per day for two weeks.
  Intervention: Behavioral - Home-based Arm and Hand Exercise
  Interventions: Behavioral: Home-based Arm and Hand Exercise

INTERVENTIONS:
Other: Wrist Alarm — Wrist device with alarm timer
  Arms: Treatment (Alarm Active)
Behavioral: Home-based Arm and Hand Exercise — Repeated visuomotor tasks, unilateral arm and hand movements, bilateral arm and hand movements

SUMMARY:
The purpose of this study is to find out whether the Home-based Arm and Hand Exercise (HAHE) program improves functions of the upper limb that is affected after traumatic brain injury. HAHE is made up of exercises that simulate real-life tasks.

DETAILED DESCRIPTION:
Arm and hand dysfunction, although not widely recognized, is a common and devastating consequence of traumatic brain injury (TBI). Recommendations have been published that encourage clinicians to include upper extremity retraining within the TBI population; however, very little research exists that will help inform treatments for this population. There is urgency to broaden the scientific evidence critical to informing upper limb rehabilitation for TBI survivors. The proposed study will do just that by using a task-specific visuomotor exercise protocol that emphasizes upper limb movements which can be practiced by patients in their homes. This new home-based arm and hand exercise (HAHE) protocol is expected to improve functional recovery and quality of life among individuals with chronic upper limb impairment after moderate-to-severe TBI.

ELIGIBILITY:
Inclusion Criteria:

* Time post injury: >12 Months
* Moderate to severe TBI, with one of the following (as confirmed by medical records):

  1. Post-traumatic amnesia for over 24 hours
  2. Trauma-related intracranial neuroimaging abnormalities (based on radiology reports of the head CT scan acquired acutely)
  3. Loss of consciousness for over 30 minutes
  4. Score of over 13 on the Glasgow Coma Scale (recorded in emergency dept, but not valid if patient was intubated, sedated or intoxicated)
* Has emerged from post-traumatic amnesia (as indicated by review of medical history documents)
* Cognitively oriented (score above 23 on the Mini Mental State Examination)
* One upper limb is more affected than the other, and participant reports impaired upper limb function because of the more affected limb
* The more affected limb is at Stage 3, 4 or 5 of Arm Recovery
* Be able to complete the sequence of the HAHE protocol independently, safely and accurately by the end of the therapist-guided training

Exclusion Criteria:

* < 18 years old at the time of injury
* A history of previous neurological disorder such as stroke, seizure, multiple sclerosis, spinal cord injury, cerebral palsy, Parkinson's disease, or Alzheimer's disease. This is to assure that participants' deficits are secondary to TBI only.
* A history of significant psychiatric disorder such as schizophrenia, bipolar disorder, or obsessive-compulsive disorder. There may be potential cognitive changes due to such history, which may affect the ability in following the treatment protocol.
* A history of substance abuse requiring inpatient treatment. There may be potential cognitive changes due to such history, which may affect the ability in following the treatment protocol.
* The more affected limb is at the Stage 1, 2, 6, or 7 of Arm Recovery (Figure 2).
* Pain in the upper extremity during the upper limb function screening
* Active subluxation of the shoulders (i.e., the glenohumeral joint)
* Undergoing treatment for spasticity in the upper limb (e.g. botulinum toxin injection)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test - Functional Ability Scale (WMFT-FAS) | Week 7
  Measures upper extremity motor ability through 15 timed and functional tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Peii Chen, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States